CLINICAL TRIAL: NCT04532047
Title: PEARL (PrEnAtal Enzyme Replacement Therapy for Lysosomal Storage Disorders)
Acronym: PEARL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Tippi Mackenzie, Professor of Surgery, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-31520
Record Dates: First submitted 2020-08-19; First posted 2020-08-31 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: MPS I; MPS II; MPS IVA; MPS VI; Mps VII; Gaucher Disease, Type 2; Gaucher Disease, Type 3; Pompe Disease Infantile-Onset; Wolman Disease
MeSH Terms: conditions — Sudden Infant Death; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Gaucher Disease; Wolman Disease | interventions — Iduronidase; idursulfase; GALNS protein, human; galsulfase; vestronidase alfa; GAA protein, human; Sebelipase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: in utero enzyme replacement therapy (Experimental): ERT will be delivered in utero. Typically, the target of the procedure to administer in utero ERT will be the umbilical vein near the insertion of the umbilical cord into the placenta. The dose of the ERT will be dependent on the specific disease process and enzyme being replaced, and the estimated weight of the fetus. The dosage will be the same as the recommended weight-based postnatal dosing, adjusted for estimated fetal weight. IUERT will be repeated every 2-4 weeks, which is an interval consistent with the standard of care for IUTs (every 2-4 weeks) to avoid excessive access through the umbilical vein. This interval is also consistent with the half-life of each relevant enzyme.
  Interventions: Drug: Aldurazyme (laronidase)

INTERVENTIONS:
Drug: Aldurazyme (laronidase) — Enzyme replacement therapy for lysosomal storage diseases
  Other Names: Elaprase (idursulfase); Vimizim (elosulfase alfa); Naglazyme (galsulfase); Mepsevii (vestronidase alfa-vjbk); Lumizyme (alglucosidase alfa); Kanuma (sebelipase alfa)

SUMMARY:
For detailed information, please view our study website: https://pearltrial.ucsf.edu/

The investigators aims to determine the the maternal and fetal safety and feasibility of in utero fetal enzyme replacement therapy in fetuses with Lysosomal Storage Diseases.

DETAILED DESCRIPTION:
Because fetuses with these LSDs are at increased risk of serious perinatal morbidity and mortality, particularly in the setting of Non-Immune Hydrops Fetalis (NIHF), the administration of the approved enzyme therapy in utero has the potential to significantly improve outcomes for affected fetuses. The perinatal death rate associated with NIHF ranges from 30 to 75%, so development of an in utero approach to treatment could be of significant benefit. The in utero period has been shown to be a time of relative fetal tolerance to immune stimuli, and this tolerance may lead to improved response to ERT in situations where postnatal initiation instead leads to antibody development and impaired response to treatment. It is also probable that in some cases, initiation of ERT in utero leads to improved neurodevelopmental outcomes if the replaced enzyme impacts the neurologic system during critical periods of development.

This is a phase 1 clinical trial to determine the safety and feasibility of fetal enzyme replacement therapy in fetuses with LSD

ELIGIBILITY:
Inclusion Criteria:

* Live male or female fetuses at 18 0/7 weeks to 34 6/7 weeks gestation
* Diagnosis of one of the 8 included LSDs in utero by genetic or enzymatic analyses performed on amniotic fluid, fetal blood, placental tissue, or other samples through chorionic villus sampling (CVS), amniocentesis, cordocentesis, cell free fetal DNA, or other procedures. In the event that parents are identified as genetic carriers for a LSD, diagnostic testing for the fetus would be performed to confirm the diagnosis
* Pregnant women age 18 years to 50 years, carrying a live male or female fetus at 18 0/7 weeks to 34 6/7 weeks gestation
* Identified through the above listed means to be carrying a fetus with an LSD.
* Ability to give written informed consent and comply with the requirements of the study.

Exclusion Criteria:

* Fetuses with a concurrent severe structural anomaly
* Fetuses with an additional pathogenic genetic variant not related to the underlying LSD that contribute a significant risk of morbidity or mortality.

Hydrops fetalis will not be an exclusion criterion because ERT has the possibility of significant benefit in this situation.

* Women with one or more significant comorbidities that would preclude fetal intervention including, but not limited to:

  1. inability to complete the procedure secondary to maternal body habitus or placental location
  2. significant cardiopulmonary disease
  3. mirror syndrome
  4. end organ failure
  5. altered mental status
  6. placental abruption
  7. active preterm labor
  8. preterm premature rupture of membranes.
* Mother will require therapeutic dosing of anticoagulation within 24 hours prior to or following the intervention.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Maternal pregnant women of age 18-50, carrying a male or female fetus at 18 0/7 weeks to 34 6/7 weeks.
Enrollment: 10 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | 6 years
  Adverse and serious adverse events including, but not limited to, death within 24 hours after the procedure, stillbirth, death prior to initial hospital discharge,increased response with antibody development above that expected with postnatal ERT, and serious related or serious unexpected adverse events exceeding those expected with the natural history of treated disease during the first five years of life, assessed by CTCAE v5.0.
Number of participants to receive the full initial, weight-based dose of enzyme replacement therapy through the fetal umbilical vein, and subsequent doses throughout the pregnancy. | 6 years
  full dose administration compared to the need to halt the intervention prior to administration of a full dose.
Number of participants with the presence and levels of glycosaminoglycans (GAGs) in urine. | 6 years
  Laboratory analysis of urine for GAG levels.
The number of participants with improvement or resolution of hydrops (if present). | 6 years
  Improvement of hydrops via ultrasound and echocardiogram results (if present).

SECONDARY OUTCOMES:
Number of participants that show measured levels of antibodies against the enzyme. | 6 years
  Laboratory analysis of blood to measure antibody levels.

OTHER OUTCOMES:
Number of participants that show functional cardiac, growth, mobility, and neurocognitive function. | 6 years
  ecogardiogram, skeletal survey, neurocognitve assessments such as Bayley III to assess cardiac, growth, mobility and neurocognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Tippi MacKenzie, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen QH, Witt RG, Wang B, Eikani C, Shea J, Smith LK, Boyle G, Cadaoas J, Sper R, MacKenzie JD, Villeda S, MacKenzie TC. Tolerance induction and microglial engraftment after fetal therapy without conditioning in mice with Mucopolysaccharidosis type VII. Sci Transl Med. 2020 Feb 26;12(532):eaay8980. doi: 10.1126/scitranslmed.aay8980. PMID 32102934
- [Background] Platt FM, d'Azzo A, Davidson BL, Neufeld EF, Tifft CJ. Author Correction: Lysosomal storage diseases. Nat Rev Dis Primers. 2018 Oct 18;4(1):36. doi: 10.1038/s41572-018-0037-0. PMID 30337566
- [Background] Meikle PJ, Hopwood JJ, Clague AE, Carey WF. Prevalence of lysosomal storage disorders. JAMA. 1999 Jan 20;281(3):249-54. doi: 10.1001/jama.281.3.249. PMID 9918480
- [Background] Azevedo AC, Schwartz IV, Kalakun L, Brustolin S, Burin MG, Beheregaray AP, Leistner S, Giugliani C, Rosa M, Barrios P, Marinho D, Esteves P, Valadares E, Boy R, Horovitz D, Mabe P, da Silva LC, de Souza IC, Ribeiro M, Martins AM, Palhares D, Kim CA, Giugliani R. Clinical and biochemical study of 28 patients with mucopolysaccharidosis type VI. Clin Genet. 2004 Sep;66(3):208-13. doi: 10.1111/j.1399-0004.2004.00277.x. PMID 15324318
- [Background] Rosenbloom BE, Weinreb NJ. Gaucher disease: a comprehensive review. Crit Rev Oncog. 2013;18(3):163-75. doi: 10.1615/critrevoncog.2013006060. PMID 23510062
- [Background] Chien YH, Lee NC, Thurberg BL, Chiang SC, Zhang XK, Keutzer J, Huang AC, Wu MH, Huang PH, Tsai FJ, Chen YT, Hwu WL. Pompe disease in infants: improving the prognosis by newborn screening and early treatment. Pediatrics. 2009 Dec;124(6):e1116-25. doi: 10.1542/peds.2008-3667. PMID 19948615
- [Background] Blitz MJ, Rochelson B, Sood M, Bialer MG, Vohra N. Prenatal sonographic findings in a case of Wolman's disease. J Clin Ultrasound. 2018 Jan;46(1):66-68. doi: 10.1002/jcu.22481. Epub 2017 Apr 4. PMID 28374935
- [Background] Tsai AC, Hung YW, Harding C, Koeller DM, Wang J, Wong LC. Next generation deep sequencing corrects diagnostic pitfalls of traditional molecular approach in a patient with prenatal onset of Pompe disease. Am J Med Genet A. 2017 Sep;173(9):2500-2504. doi: 10.1002/ajmg.a.38333. Epub 2017 Jun 28. PMID 28657663
- [Background] Banugaria SG, Prater SN, Ng YK, Kobori JA, Finkel RS, Ladda RL, Chen YT, Rosenberg AS, Kishnani PS. The impact of antibodies on clinical outcomes in diseases treated with therapeutic protein: lessons learned from infantile Pompe disease. Genet Med. 2011 Aug;13(8):729-36. doi: 10.1097/GIM.0b013e3182174703. PMID 21637107
- [Derived] Borges B, Canepa E, Chang IJ, Herzeg A, Lianoglou B, Kishnani PS, Harmatz P, MacKenzie TC, Cohen JL. Prenatal Delivery of Enzyme Replacement Therapy to Fetuses Affected by Early-Onset Lysosomal Storage Diseases. Am J Med Genet C Semin Med Genet. 2025 Sep;199(3):203-217. doi: 10.1002/ajmg.c.32132. Epub 2025 Jan 31. PMID 39891377
- [Derived] Herzeg A, Borges B, Lianoglou BR, Gonzalez-Velez J, Canepa E, Munar D, Young SP, Bali D, Gelb MH, Chakraborty P, Kishnani PS, Harmatz P, Cohen JL, MacKenzie TC. Intrauterine enzyme replacement therapies for lysosomal storage disorders: Current developments and promising future prospects. Prenat Diagn. 2023 Dec;43(13):1638-1649. doi: 10.1002/pd.6460. Epub 2023 Nov 13. PMID 37955580